CLINICAL TRIAL: NCT06661681
Title: Cognitive Functional Therapy Versus Therapeutic Exercises for the Treatment of Individuals With Chronic Shoulder Pain: A Randomized Controlled Trial
Brief Title: Cognitive Functional Therapy for Treating Individuals With Chronic Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Danilo Harudy Kamonseki, Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 409730/2023-8
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Shoulder Pain; Exercise Therapy; Psychosocial Rehabilitation
Keywords: Shoulder pain; Subacromial pain; Rotator cuff related shoulder pain; Shoulder Impingement; Chronic pain; Psychosocial; Rehabilitation; Biopsychosocial
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a superiority randomized controlled trial, single-blinded, with two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: Evaluators will be blinded to the treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Functional Therapy (Experimental): Cognitive Functional Therapy (CFT) will be conducted weekly in sessions lasting approximately 60 minutes over 8 weeks.
  Interventions: Behavioral: Cognitive Functional Therapy (CFT)
- Therapeutic exercises group (Active Comparator): Individuals assigned to this group will be treated twice a week for eight weeks, wich each session will last approximately 40 to 60 minutes.
  Interventions: Other: Therapeutic exercises group

INTERVENTIONS:
Behavioral: Cognitive Functional Therapy (CFT) — Cognitive Functional Therapy (CFT) is underpinned by a strong therapeutic alliance, active listening, and motivational interviewing style, covering the following domains:
  i) Making sense of pain involves discussing the multidimensional nature of persistent pain, as well as the beliefs, emotions, and behaviors that can perpetuate the vicious cycle of pain and disability.
  ii) Exposure with control involves a functional training designed to normalize maladaptive and provocative postural and movement behaviors, where individuals will learn strategies to improve their body awareness and control and modify postures and tasks commonly associated with pain.
  iii) Lifestyle change aims to help patients embrace a healthy lifestyle, which will include promoting a gradual increase in physical activity, sleep hygiene counseling, stress management strategies, and social re-engagement.
  Other Names: CFT
  Arms: Cognitive Functional Therapy
Other: Therapeutic exercises group — Each session will include stretching exercises targeting the following muscles i) Upper trapezius; ii) Pectoralis minor; iii) Posterior shoulder region, and strengthening exercises targeting the following muscles i) Lower trapezius, ii) Middle trapezius, iii) Serratus punch exercise, iv) Shoulder external rotators, and v) Shoulder internal rotators.
  Arms: Therapeutic exercises group

SUMMARY:
Shoulder pain is a debilitating musculoskeletal condition with functional, physical, and psychological impacts. Interventions for chronic shoulder pain should address the biopsychosocial model, with Cognitive Functional Therapy emerging as a promising physiotherapy approach. Cognitive Functional Therapy approaches the multidimensional nature of pain, integrating physical and cognitive aspects.

The aim of this randomized controlled trial is to compare the effects of Cognitive Functional Therapy with therapeutic exercise on biological aspects of pain (pain intensity, disability, function, perception of improvement/deterioration, and central pain processing), and psychosocial aspects of pain (sleep quality, self-efficacy, and biopsychosocial factors). The hypothesis of this study is that CFT will lead to greater improvements in these outcomes compared to therapeutic exercise.

DETAILED DESCRIPTION:
This will be a randomized controlled trial, single-blinded with two parallel groups. Seventy-two individuals with chronic shoulder pain will be randomly assigned to one of two groups: CFT or Therapeutic exercises. The interventions will last eight weeks, with the CFT group receiving therapy once a week and the therapeutic exercise group receiving sessions twice weekly. The primary outcomes will be pain intensity and disability, while the secondary outcomes will include function, self-efficacy, sleep quality, biopsychosocial factors, perception of improvement/deterioration, and central pain processing.

ELIGIBILITY:
Inclusion Criteria:

* Men or women;
* Age between 18 and 60 years;
* Presence of shoulder pain for more than 3 months;
* Pain intensity of 4 points or more on the 11-point Numeric Pain Rating Scale.
* High level of disability or moderate level of irritability.

Exclusion Criteria:

* History of fracture or surgery of the clavicle, scapula, and/or humerus, surgical stabilization or rotator cuff repair;
* History of dislocation, instability (positive sulcus sign or apprehension test), and/or rotator cuff tear (positive drop arm test);
* Adhesive capsulitis verified by the presence of gradual onset pain associated with stiffness and reduced passive and active mobility;
* Ongoing pregnancy;
* Reproduction of shoulder pain radiating to the entire upper limb during cervical or thoracic spine tests (positive Spurling test);
* Neurological or systemic diseases that may alter muscle strength and sensitivity such as rheumatoid arthritis, fibromyalgia, lupus, gout, and diabetes;
* Corticosteroid injection in the shoulder region in the last 3 months;
* Physiotherapy treatment in the last 6 months.
* Active treatment for cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Pain intensity: Numerical Pain Rating Scale (NPRS) | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  The pain intensity will be measured with 11 point - Numerical Rating Pain Scale (NPRS) with scores ranging from 0 (no pain) to 10 (maximum pain). Higher scores indicate greater pain intensity.
Disability: Shoulder Pain and Disability Index (SPADI) | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Disability will be assessed with Shoulder Pain and Disability Index (SPADI). which is composed of 13 questions related to two domains: disability (eight items) and pain (five items). The final score ranges from 0 to 100, with higher scores indicating greater shoulder disability

SECONDARY OUTCOMES:
Shoulder function: Patient Specific Functional Scale | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Shoulder functional ability will be measured with Patient Specific Functional Scale. The individuals will select three to five important activities that are challenging to perform due to shoulder pain. For each reported activity, the individual will score on an 11-point scale, where 0 is (unable to perform the activity) and 10 is (able to perform the activity at the level prior to the injury). Score ranges from 0 (unable to perform) to 10 (able to perform at preinjury level). Higher score means better function.
Self-efficacy: Pain Self-Efficacy Questionnaire (PSEQ) | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Self-efficacy will be assessed with Pain Self-Efficacy Questionnaire (PSEQ) will be used to assess, which is composed of of 10 items. The total score ranges from 0 to 60 points, with the higher score indicating greater self-efficacy.
Sleep quality: Pittsburgh Sleep Quality Index (PSQI) | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Sleep quality will be assessed with Pittsburgh Sleep Quality Index (PSQI), which is composed of 19 items, resulting in a total score ranging from 0 to 21, and covering 7 domains: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbance, (6) medication use and (7) dysfunction during the day. The total score ranges from 0 to 21, with higher scores indicating worse sleep quality.
Biopsychosocial Aspects: Brief Screening Questions for Biopsychosocial Aspects | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Biopsychosocial Aspects will be assessed with the Brief Screening Questions for Biopsychosocial, which is composed of six questions covering five domains: anxiety, kinesiophobia, stress, catastrophizing, and depression. The scores for each question range from 0 to 10, with higher scores indicating worse symptoms.
Perception of improvement/deterioration over time: Global Rating of Change Scale | 4-week, at the end of treatment (8-week), and 12-week follow-up
  The individual's perception of improvement/deterioration over time will be measured with the Global Rating of Change Scale, which ranges from -7 to 7, with positive and higher scores indicating a greater perception of health improvement, negative and lower scores indicating a worsening perception of health, and a score of zero representing no change.
Central pain processing: Pressure Pain Threshold (PPT) | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Pressure Pain Threshold (PPT) is defined as the minimum amount of pressure that triggers the first sensation of pain. Pressure Pain Threshold will be measured by a digital pressure algometer (AlgoMed ®, Hӧrby, Sweden) with 1 cm2 circular rubber probe tip and a pressure rate of approximately 40 kPa/s. The Pressure Pain Threshold test will be performed at the acromion and muscle bellies of the deltoid, upper trapezius, and tibialis anterior.
Central pain processing: Temporal summation | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Temporal summation refers to increased perceived pain from repetitive nociceptive stimuli at the same site, which is related to the modulation mechanism occurring in second-order sensory neurons in the spinal cord. The temporal summation will be measured at the deltoid and tibialis anterior. Sequential stimulation will involve 10 pressure stimuli at the pre-established Pressure Pain Threshold level, with a one-second interval between stimuli. Each pressure increment will be approximately 40 kPa/s. After the first and tenth stimuli, participants will rate their pain intensity using the Numerical Rating Pain Scale (NPRS) with scores ranging from 0 (no pain) to 10 (maximum pain), and higher scores indicate greater pain intensity. The temporal summation will be quantified by subtracting the pain intensity rating for the first stimulus from the pain rating for the tenth.
Central pain processing: Conditioned Pain Modulation | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Conditioned Pain Modulation (CPM) refers to the central nervous system's ability to inhibit pain through mechanisms related to endogenous descending inhibition. Individuals will immerse their hand in a cold-water bath for 2 minutes. Pressure Pain Threshold (PPT) at the deltoid of the affected (or most affected) side will be assessed at baseline, during immersion (after 30, 60, and 90 seconds), and after immersion (immediately post-withdrawal and at 30 and 60 seconds after withdrawal). Participants will rate their pain intensity on the Numerical Rating Pain Scale (NPRS) with scores ranging from 0 (no pain) to 10 (maximum pain), and higher scores indicate greater pain intensity, every 30 seconds from immersion until hand withdrawal, and 30 and 60 seconds after withdrawal. CPM will be calculated by subtracting the PPT of the deltoid from PPT measures during and after Conditioned Pain Modulation.

CONTACTS AND LOCATIONS:
Overall Officials: Danilo H Kamonseki, PhD, Principal Investigator — Universidade Federal da Paraíba
Locations (1):
- Federal University of Paraíba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared under request.
Supporting Information: Study Protocol, SAP
Time Frame: baseline, 4th week, end of treatment (8th week), and 12th-week follow-up.